CLINICAL TRIAL: NCT05218603
Title: A Prospective, Observational Study, to Evaluate the Maintenance With Bortezomib Plus Daratumumab (V-Dara) After Induction With Bortezomib, Melphalan, Prednisone Plus Daratumumab (VMP-Dara) in Newly Diagnosed Multiple Myeloma (MM) Patients Non-eligible for Autologous Stem Cell Transplantation (ASCT): Alcyone-optimized Real World Evidence (RWE) Data
Brief Title: Evaluation of Maintenance With Bortezomib Plus Daratumumab (V-Dara) After Induction With Bortezomib, Melphalan, Prednisone Plus Daratumumab (VMP-Dara) in Newly Diagnosed Multiple Myeloma (MM) Patients Non-eligible for autoSCT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: PETHEMA Foundation (Other)
Collaborators: Janssen, LP (Industry); Adknoma Health Research (Industry)
Responsible Party: Sponsor
Other Study IDs: GEM-OPTIMAL
Record Dates: First submitted 2022-01-17; First posted 2022-02-01 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: Multiple Myeloma; Non-eligible for Autologous Stem Cell Transplantation (ASCT)
Keywords: Prospective; Observational study; Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib; daratumumab

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Maintenance with V-Dara after receiving VMP-Dara as induction regimen: Maintenance with bortezomib plus daratumumab (V-Dara) after induction with bortezomib, melphalan, prednisone plus daratumumab (VMP-Dara)
  Interventions: Drug: Bortezomib; Drug: Daratumumab

INTERVENTIONS:
Drug: Bortezomib — Maintenance: Administration as per routine clinical practice.
Drug: Daratumumab — Maintenance: Administration as per routine clinical practice.

SUMMARY:
This is a prospective, observational, single group and multicenter study to describe the effectiveness and safety of maintenance with V-Dara after induction with the VMP-Dara regimen in newly diagnosed MM patients who are not eligible for ASCT.

Patients will be enrolled in the study during a regularly scheduled office visit in clinical practice (screening and enrollment visit) and followed during 3-4 years in what will be called the Observational Phase. During this phase, the patient will be followed by his/her doctor as per routine clinical practice, according to his/her disease. The patient will not suffer any changes in his/her treatment or follow-up due to his/her participation in the study. The patient will receive standard clinical practice and he/she will not do any other study-specific visit.

During this 3-4-year observational phase, the patient might discontinue V or V-Dara,depending on toxicity, efficacy or due to other medical reasons, according to his/her physician decision.

DETAILED DESCRIPTION:
This is a prospective, observational, single group and multicenter study to describe the effectiveness and safety of maintenance with V-Dara after induction with the VMP-Dara regimen in newly diagnosed MM patients who are not eligible for ASCT.

Patients will be recruited only if patients have received induction therapy with VMP-Dara followed by V-Dara as maintenance therapy for at least one cycle prior to the start of the study (treatment has to be previously decided as part of clinical practice). This way, patients must have already been treated with 9 cycles of VMP-Dara (approximately 12 months) and at least 1 cycle of V-Dara maintenance (1 month), before entering the study. This implies that the decision to prescribe this maintenance schedule is clearly unrelated to the decision of enrolling the patient into the study.

Patients will be enrolled in the study during a regularly scheduled office visit in clinical practice (screening and enrollment visit) and followed during 3-4 years in what will be called the Observational Phase. During this phase, the patient will be followed by his/her doctor as per routine clinical practice, according to his/her disease. The patient will not suffer any changes in his/her treatment or follow-up due to his/her participation in the study. The patient will receive standard clinical practice and he/she will not do any other study-specific visit.

Observational Phase:

Patients will be followed for 3-4 years since the inclusion in the study. Once the patient is enrolled in the study, retrospective data collection at the start and end of VMP-Dara induction will be collected. Subjects who discontinue maintenance therapy before disease progression (V or V-Dara), will continue to have response rate evaluations, PFS and toxicity recorded as per routine clinical practice, until the end of the study or progression, whatever comes first.

During this observational follow-up, both the duration of the initially prescribed V-Dara maintenance (and the time when bortezomib is stopped before daratumumab if this ever happens), the existence of potential adverse reactions and the fate of the disease in terms of progression and survival, even though the maintenance only daratumumab could have been stopped, will be documented for a total of up to 3-4 years. Maintenance with V-Dara, or just daratumumab once bortezomib is suspended, can be finalized due to progression, unacceptable toxicity or voluntary withdrawal.

This observational study has the following objectives:

Primary Objective:

- To describe the effectiveness of V-Dara maintenance after VMPDara induction in patients with MM non-eligible for autologous stem cell transplantation in the Spanish clinical setting (clinical practice).

Secondary Objectives:

* Compare the effectiveness of VMP-Dara induction followed by V-Dara maintenance with the results of the Daratumumab arm of the Alcyone trial (VMP-Dara followed by Dara maintenance).
* To describe the safety of the V-Dara maintenance therapy used in clinical practice after VMP-Dara.
* To evaluate the clinical effectiveness in different risk subgroups.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a newly diagnosed MM non eligible for ASCT that have received induction therapy with D-VMP (9 cycles) and followed by V-Dara as maintenance* in clinical practice. The decision to prescribe maintenance treatment with V-Dara must be in accordance with clinical practice, must not be influenced by the planned inclusion of a patient in the study, and should be documented before enrollment.
2. Patients ≥18 years of age.
3. Each subject (or their legally acceptable representative) must sign the ICF indicating that he or she understands the purpose of the observational nature the study and are willing to share his/her clinical data for the study.

Exclusion Criteria:

1. Patients with a diagnosis of primary amyloidosis, monoclonal gammopathy of undetermined significance, smoldering MM, plasma cell leukemia, POEMS syndrome, Waldenström's disease, or other conditions in which IgM M-protein is present in the absence of a clonal plasma cell infiltration with lytic bone lesions.
2. Subjects with prior or current systemic therapy or ASCT for MM (before VMP-Dara induction), except for an emergency use of a short course of corticosteroids before treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A target of approximately 100 subjects from the centers opened in the study will be recruited only if patients have received induction therapy with VMP-Dara followed by V-Dara as maintenance therapy for at least one cycle prior to the start of the study (treatment has to be previously decided as part of clinical practice). This way, patients must have already been treated with 9 cycles of VMP-Dara (approximately 12 months) and at least 1 cycle of V-Dara maintenance (1 month), before entering the study. This implies that the decision to prescribe this maintenance schedule is clearly unrelated to the decision of enrolling the patient into the study.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-11-30 (Actual); Primary Completion 2025-11-06 (Estimated); Study Completion 2025-11-06 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | Throughout the study period. Approximately 4 years
  Time from the start of induction with VMPDara until disease progression or death, whichever comes first

SECONDARY OUTCOMES:
Description of MRD status and depth | Throughout the study period. Approximately 4 years
  Description of MRD status and depth, that will be conducted on bone marrow samples and outside of the bone marrow through imaging techniques if available per routine clinical practice, according to the investigator's criteria.
Stringent Complete Response (sCR) rate | Throughout the study period. Approximately 4 years
Complete Response (CR) rate | Throughout the study period. Approximately 4 years
Proportion of subjects who achieve Very Good Partial Response (VGPR) or better | Throughout the study period. Approximately 4 years
Overall Response Rate (ORR) | Throughout the study period. Approximately 4 years
Duration of response | Throughout the study period. Approximately 4 years
  Duration of response calculated from the date of initial documentation of a response (CR or PR) to the date of first documented evidence of progressive disease.
Time to Progression (TTP) | Throughout the study period. Approximately 4 years
  Time to Progression (TTP), defined as the time from the date of start of VMP-Dara to the date of first documented evidence of PD.
Incidence of adverse events (AEs) | Throughout the study period. Approximately 4 years
  Number of patients experiencing AEs, classified according to severity.

CONTACTS AND LOCATIONS:
Overall Officials: María Victoria Mateos Manteca, Principal Investigator — Hospital Universitario de Salamanca (Salamanca); Jesús San Miguel Izquierdo, Principal Investigator — Clínica Universidad de Navarra (Pamplona)
Locations (32):
- Spain (32):
  - Hospital Universitario Del Sureste, Arganda
  - Complejo Asistencial de Avila, Ávila
  - Hospital Quirón Sagrado Corazón, Barcelona
  - Hsopital Clinic de Barcelona, Barcelona
  - Hospital Universitario Virgen de Las Nieves, Granada
  - Complejo Hospitalario de Jaén, Jaén
  - Complejo Hospitalario Universitario de Gran Canaria Dr. Negrín, Las Palmas de Gran Canaria
  - Hospital de León, León
  - Hospital Clínico San Carlos, Madrid
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Ramón Y Cajal, Madrid
  - Hospital Ruber Juan Bravo 39, Madrid
  - Hospital Universitario de La Princesa, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital Universitario Infanta Leonor, Madrid
  - Hospital General Universitario J.M. Morales Meseguer, Murcia
  - Complexo Hospitalario Universitario de Ourense, Ourense
  - Hospital Universitario Central de Asturias, Oviedo
  - Clinica Universidad de Navarra, Pamplona
  - Hospital Virgen Del Puerto, Plasencia
  - Hospital El Bierzo, Ponferrada
  - Hospital Montecelo, Pontevedra
  - Hospital Quirónsalud Madrid, Pozuelo de Alarcón
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Universitario de Canarias (H.U.C), San Cristóbal de La Laguna
  - Hospital Universitario Infanta Sofía, San Sebastián de los Reyes
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Hospital Clinico Universitario de Santiago, Santiago de Compostela
  - Hospital General Nuestra Señora Del Prado, Talavera de la Reina
  - Hospital Universitari Mútua de Terrassa, Terrassa
  - Hospital General de Tomelloso, Tomelloso
  - Hospital Clinico Universitario de Valladolid, Valladolid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Palumbo A, Anderson K. Multiple myeloma. N Engl J Med. 2011 Mar 17;364(11):1046-60. doi: 10.1056/NEJMra1011442. No abstract available. PMID 21410373
- [Background] Jemal A, Siegel R, Xu J, Ward E. Cancer statistics, 2010. CA Cancer J Clin. 2010 Sep-Oct;60(5):277-300. doi: 10.3322/caac.20073. Epub 2010 Jul 7. PMID 20610543
- [Background] Al-Farsi K. Multiple myeloma: an update. Oman Med J. 2013 Jan;28(1):3-11. doi: 10.5001/omj.2013.02. PMID 23386937
- [Background] Bianchi G, Richardson PG, Anderson KC. Promising therapies in multiple myeloma. Blood. 2015 Jul 16;126(3):300-10. doi: 10.1182/blood-2015-03-575365. Epub 2015 Jun 1. No abstract available. PMID 26031917
- [Background] Anderson KC. Progress and Paradigms in Multiple Myeloma. Clin Cancer Res. 2016 Nov 15;22(22):5419-5427. doi: 10.1158/1078-0432.CCR-16-0625. PMID 28151709
- [Background] Kumar SK, Rajkumar V, Kyle RA, van Duin M, Sonneveld P, Mateos MV, Gay F, Anderson KC. Multiple myeloma. Nat Rev Dis Primers. 2017 Jul 20;3:17046. doi: 10.1038/nrdp.2017.46. PMID 28726797
- [Background] Mihelic R, Kaufman JL, Lonial S. Maintenance therapy in multiple myeloma. Leukemia. 2007 Jun;21(6):1150-7. doi: 10.1038/sj.leu.2404633. Epub 2007 Mar 8. PMID 17344913
- [Background] Ludwig H, Durie BG, McCarthy P, Palumbo A, San Miguel J, Barlogie B, Morgan G, Sonneveld P, Spencer A, Andersen KC, Facon T, Stewart KA, Einsele H, Mateos MV, Wijermans P, Waage A, Beksac M, Richardson PG, Hulin C, Niesvizky R, Lokhorst H, Landgren O, Bergsagel PL, Orlowski R, Hinke A, Cavo M, Attal M; International Myeloma Working Group. IMWG consensus on maintenance therapy in multiple myeloma. Blood. 2012 Mar 29;119(13):3003-15. doi: 10.1182/blood-2011-11-374249. Epub 2012 Jan 23. PMID 22271445
- [Background] Nooka, A.K., Behera, M., Boise, L.H., Kaufman, J.L., Watson, M. and Lonial, S. (2011) Thalidomide as maintenance therapy in multiple myeloma (MM) improves progression free survival (PFS) and overall survival (OS): a meta-analysis. ASH Annu. Meet. Abstr. 118, 1855
- [Background] Hahn, A., Lilienfeld, T.M. and Heteren, P. (2011) Improved progression-free and overall survival with thalidomide maintenance therapy after autologous stem cell transplantation in multiple myeloma: a meta-analysis of five randomized trials. Haematologica 96, 884.
- [Background] Morgan GJ, Gregory WM, Davies FE, Bell SE, Szubert AJ, Brown JM, Coy NN, Cook G, Russell NH, Rudin C, Roddie H, Drayson MT, Owen RG, Ross FM, Jackson GH, Child JA; National Cancer Research Institute Haematological Oncology Clinical Studies Group. The role of maintenance thalidomide therapy in multiple myeloma: MRC Myeloma IX results and meta-analysis. Blood. 2012 Jan 5;119(1):7-15. doi: 10.1182/blood-2011-06-357038. Epub 2011 Oct 20. PMID 22021371
- [Background] Palumbo A, Bringhen S, Caravita T, Merla E, Capparella V, Callea V, Cangialosi C, Grasso M, Rossini F, Galli M, Catalano L, Zamagni E, Petrucci MT, De Stefano V, Ceccarelli M, Ambrosini MT, Avonto I, Falco P, Ciccone G, Liberati AM, Musto P, Boccadoro M; Italian Multiple Myeloma Network, GIMEMA. Oral melphalan and prednisone chemotherapy plus thalidomide compared with melphalan and prednisone alone in elderly patients with multiple myeloma: randomised controlled trial. Lancet. 2006 Mar 11;367(9513):825-31. doi: 10.1016/S0140-6736(06)68338-4. PMID 16530576
- [Background] Wijermans P, Schaafsma M, Termorshuizen F, Ammerlaan R, Wittebol S, Sinnige H, Zweegman S, van Marwijk Kooy M, van der Griend R, Lokhorst H, Sonneveld P; Dutch-Belgium Cooperative Group HOVON. Phase III study of the value of thalidomide added to melphalan plus prednisone in elderly patients with newly diagnosed multiple myeloma: the HOVON 49 Study. J Clin Oncol. 2010 Jul 1;28(19):3160-6. doi: 10.1200/JCO.2009.26.1610. Epub 2010 Jun 1. PMID 20516439
- [Background] Waage A, Gimsing P, Fayers P, Abildgaard N, Ahlberg L, Bjorkstrand B, Carlson K, Dahl IM, Forsberg K, Gulbrandsen N, Haukas E, Hjertner O, Hjorth M, Karlsson T, Knudsen LM, Nielsen JL, Linder O, Mellqvist UH, Nesthus I, Rolke J, Strandberg M, Sorbo JH, Wisloff F, Juliusson G, Turesson I; Nordic Myeloma Study Group. Melphalan and prednisone plus thalidomide or placebo in elderly patients with multiple myeloma. Blood. 2010 Sep 2;116(9):1405-12. doi: 10.1182/blood-2009-08-237974. Epub 2010 May 6. PMID 20448107
- [Background] Beksac M, Haznedar R, Firatli-Tuglular T, Ozdogu H, Aydogdu I, Konuk N, Sucak G, Kaygusuz I, Karakus S, Kaya E, Ali R, Gulbas Z, Ozet G, Goker H, Undar L. Addition of thalidomide to oral melphalan/prednisone in patients with multiple myeloma not eligible for transplantation: results of a randomized trial from the Turkish Myeloma Study Group. Eur J Haematol. 2011 Jan;86(1):16-22. doi: 10.1111/j.1600-0609.2010.01524.x. Epub 2010 Nov 22. PMID 20942865
- [Background] Yang B, Yu RL, Chi XH, Lu XC. Lenalidomide treatment for multiple myeloma: systematic review and meta-analysis of randomized controlled trials. PLoS One. 2013 May 14;8(5):e64354. doi: 10.1371/journal.pone.0064354. Print 2013. PMID 23691202
- [Background] Palumbo A, Bringhen S, Kumar SK, Lupparelli G, Usmani S, Waage A, Larocca A, van der Holt B, Musto P, Offidani M, Petrucci MT, Evangelista A, Zweegman S, Nooka AK, Spencer A, Dimopoulos MA, Hajek R, Cavo M, Richardson P, Lonial S, Ciccone G, Boccadoro M, Anderson K, Barlogie B, Sonneveld P, McCarthy PL. Second primary malignancies with lenalidomide therapy for newly diagnosed myeloma: a meta-analysis of individual patient data. Lancet Oncol. 2014 Mar;15(3):333-42. doi: 10.1016/S1470-2045(13)70609-0. Epub 2014 Feb 11. PMID 24525202
- [Background] Adams J. The proteasome: a suitable antineoplastic target. Nat Rev Cancer. 2004 May;4(5):349-60. doi: 10.1038/nrc1361. No abstract available. PMID 15122206
- [Background] Yang H, Zonder JA, Dou QP. Clinical development of novel proteasome inhibitors for cancer treatment. Expert Opin Investig Drugs. 2009 Jul;18(7):957-71. doi: 10.1517/13543780903002074. PMID 19505187
- [Background] Avet-Loiseau H, Leleu X, Roussel M, Moreau P, Guerin-Charbonnel C, Caillot D, Marit G, Benboubker L, Voillat L, Mathiot C, Kolb B, Macro M, Campion L, Wetterwald M, Stoppa AM, Hulin C, Facon T, Attal M, Minvielle S, Harousseau JL. Bortezomib plus dexamethasone induction improves outcome of patients with t(4;14) myeloma but not outcome of patients with del(17p). J Clin Oncol. 2010 Oct 20;28(30):4630-4. doi: 10.1200/JCO.2010.28.3945. Epub 2010 Jul 19. PMID 20644101
- [Background] McCarthy PL, Einsele H, Attal M, Giralt S. The emerging role of consolidation and maintenance therapy for transplant-eligible multiple myeloma patients. Expert Rev Hematol. 2014 Feb;7(1):55-66. doi: 10.1586/17474086.2014.878645. Epub 2014 Jan 29. PMID 24471885
- [Background] Rollig C, Knop S, Bornhauser M. Multiple myeloma. Lancet. 2015 May 30;385(9983):2197-208. doi: 10.1016/S0140-6736(14)60493-1. Epub 2014 Dec 23. PMID 25540889
- [Background] Sun CY, Li JY, Chu ZB, Zhang L, Chen L, Hu Y. Efficacy and safety of bortezomib maintenance in patients with newly diagnosed multiple myeloma: a meta-analysis. Biosci Rep. 2017 Jul 27;37(4):BSR20170304. doi: 10.1042/BSR20170304. Print 2017 Aug 31. PMID 28706008
- [Background] Mateos MV, Oriol A, Martinez-Lopez J, Gutierrez N, Teruel AI, de Paz R, Garcia-Larana J, Bengoechea E, Martin A, Mediavilla JD, Palomera L, de Arriba F, Gonzalez Y, Hernandez JM, Sureda A, Bello JL, Bargay J, Penalver FJ, Ribera JM, Martin-Mateos ML, Garcia-Sanz R, Cibeira MT, Ramos ML, Vidriales MB, Paiva B, Montalban MA, Lahuerta JJ, Blade J, Miguel JF. Bortezomib, melphalan, and prednisone versus bortezomib, thalidomide, and prednisone as induction therapy followed by maintenance treatment with bortezomib and thalidomide versus bortezomib and prednisone in elderly patients with untreated multiple myeloma: a randomised trial. Lancet Oncol. 2010 Oct;11(10):934-41. doi: 10.1016/S1470-2045(10)70187-X. Epub 2010 Aug 23. PMID 20739218
- [Background] Mateos MV, Oriol A, Martinez-Lopez J, Gutierrez N, Teruel AI, Lopez de la Guia A, Lopez J, Bengoechea E, Perez M, Polo M, Palomera L, de Arriba F, Gonzalez Y, Hernandez JM, Granell M, Bello JL, Bargay J, Penalver FJ, Ribera JM, Martin-Mateos ML, Garcia-Sanz R, Lahuerta JJ, Blade J, San-Miguel JF. Maintenance therapy with bortezomib plus thalidomide or bortezomib plus prednisone in elderly multiple myeloma patients included in the GEM2005MAS65 trial. Blood. 2012 Sep 27;120(13):2581-8. doi: 10.1182/blood-2012-05-427815. Epub 2012 Aug 13. PMID 22889759
- [Background] Palumbo A, Bringhen S, Rossi D, Cavalli M, Larocca A, Ria R, Offidani M, Patriarca F, Nozzoli C, Guglielmelli T, Benevolo G, Callea V, Baldini L, Morabito F, Grasso M, Leonardi G, Rizzo M, Falcone AP, Gottardi D, Montefusco V, Musto P, Petrucci MT, Ciccone G, Boccadoro M. Bortezomib-melphalan-prednisone-thalidomide followed by maintenance with bortezomib-thalidomide compared with bortezomib-melphalan-prednisone for initial treatment of multiple myeloma: a randomized controlled trial. J Clin Oncol. 2010 Dec 1;28(34):5101-9. doi: 10.1200/JCO.2010.29.8216. Epub 2010 Oct 12. PMID 20940200
- [Background] Palumbo A, Bringhen S, Larocca A, Rossi D, Di Raimondo F, Magarotto V, Patriarca F, Levi A, Benevolo G, Vincelli ID, Grasso M, Franceschini L, Gottardi D, Zambello R, Montefusco V, Falcone AP, Omede P, Marasca R, Morabito F, Mina R, Guglielmelli T, Nozzoli C, Passera R, Gaidano G, Offidani M, Ria R, Petrucci MT, Musto P, Boccadoro M, Cavo M. Bortezomib-melphalan-prednisone-thalidomide followed by maintenance with bortezomib-thalidomide compared with bortezomib-melphalan-prednisone for initial treatment of multiple myeloma: updated follow-up and improved survival. J Clin Oncol. 2014 Mar 1;32(7):634-40. doi: 10.1200/JCO.2013.52.0023. Epub 2014 Jan 21. PMID 24449241
- [Background] Mateos MV, Dimopoulos MA, Cavo M, Suzuki K, Jakubowiak A, Knop S, Doyen C, Lucio P, Nagy Z, Kaplan P, Pour L, Cook M, Grosicki S, Crepaldi A, Liberati AM, Campbell P, Shelekhova T, Yoon SS, Iosava G, Fujisaki T, Garg M, Chiu C, Wang J, Carson R, Crist W, Deraedt W, Nguyen H, Qi M, San-Miguel J; ALCYONE Trial Investigators. Daratumumab plus Bortezomib, Melphalan, and Prednisone for Untreated Myeloma. N Engl J Med. 2018 Feb 8;378(6):518-528. doi: 10.1056/NEJMoa1714678. Epub 2017 Dec 12. PMID 29231133
- [Background] Mateos MV, Richardson PG, Schlag R, Khuageva NK, Dimopoulos MA, Shpilberg O, Kropff M, Spicka I, Petrucci MT, Palumbo A, Samoilova OS, Dmoszynska A, Abdulkadyrov KM, Schots R, Jiang B, Esseltine DL, Liu K, Cakana A, van de Velde H, San Miguel JF. Bortezomib plus melphalan and prednisone compared with melphalan and prednisone in previously untreated multiple myeloma: updated follow-up and impact of subsequent therapy in the phase III VISTA trial. J Clin Oncol. 2010 May 1;28(13):2259-66. doi: 10.1200/JCO.2009.26.0638. Epub 2010 Apr 5. PMID 20368561
- [Background] Rajkumar SV, Dimopoulos MA, Palumbo A, Blade J, Merlini G, Mateos MV, Kumar S, Hillengass J, Kastritis E, Richardson P, Landgren O, Paiva B, Dispenzieri A, Weiss B, LeLeu X, Zweegman S, Lonial S, Rosinol L, Zamagni E, Jagannath S, Sezer O, Kristinsson SY, Caers J, Usmani SZ, Lahuerta JJ, Johnsen HE, Beksac M, Cavo M, Goldschmidt H, Terpos E, Kyle RA, Anderson KC, Durie BG, Miguel JF. International Myeloma Working Group updated criteria for the diagnosis of multiple myeloma. Lancet Oncol. 2014 Nov;15(12):e538-48. doi: 10.1016/S1470-2045(14)70442-5. Epub 2014 Oct 26. PMID 25439696
- [Background] Durie BG, Harousseau JL, Miguel JS, Blade J, Barlogie B, Anderson K, Gertz M, Dimopoulos M, Westin J, Sonneveld P, Ludwig H, Gahrton G, Beksac M, Crowley J, Belch A, Boccadaro M, Cavo M, Turesson I, Joshua D, Vesole D, Kyle R, Alexanian R, Tricot G, Attal M, Merlini G, Powles R, Richardson P, Shimizu K, Tosi P, Morgan G, Rajkumar SV; International Myeloma Working Group. International uniform response criteria for multiple myeloma. Leukemia. 2006 Sep;20(9):1467-73. doi: 10.1038/sj.leu.2404284. Epub 2006 Jul 20. PMID 16855634
- [Background] Rajkumar SV, Harousseau JL, Durie B, Anderson KC, Dimopoulos M, Kyle R, Blade J, Richardson P, Orlowski R, Siegel D, Jagannath S, Facon T, Avet-Loiseau H, Lonial S, Palumbo A, Zonder J, Ludwig H, Vesole D, Sezer O, Munshi NC, San Miguel J; International Myeloma Workshop Consensus Panel 1. Consensus recommendations for the uniform reporting of clinical trials: report of the International Myeloma Workshop Consensus Panel 1. Blood. 2011 May 5;117(18):4691-5. doi: 10.1182/blood-2010-10-299487. Epub 2011 Feb 3. PMID 21292775
- [Background] Kumar S, Paiva B, Anderson KC, Durie B, Landgren O, Moreau P, Munshi N, Lonial S, Blade J, Mateos MV, Dimopoulos M, Kastritis E, Boccadoro M, Orlowski R, Goldschmidt H, Spencer A, Hou J, Chng WJ, Usmani SZ, Zamagni E, Shimizu K, Jagannath S, Johnsen HE, Terpos E, Reiman A, Kyle RA, Sonneveld P, Richardson PG, McCarthy P, Ludwig H, Chen W, Cavo M, Harousseau JL, Lentzsch S, Hillengass J, Palumbo A, Orfao A, Rajkumar SV, Miguel JS, Avet-Loiseau H. International Myeloma Working Group consensus criteria for response and minimal residual disease assessment in multiple myeloma. Lancet Oncol. 2016 Aug;17(8):e328-e346. doi: 10.1016/S1470-2045(16)30206-6. PMID 27511158
- [Background] Ladetto M, Bruggemann M, Monitillo L, Ferrero S, Pepin F, Drandi D, Barbero D, Palumbo A, Passera R, Boccadoro M, Ritgen M, Gokbuget N, Zheng J, Carlton V, Trautmann H, Faham M, Pott C. Next-generation sequencing and real-time quantitative PCR for minimal residual disease detection in B-cell disorders. Leukemia. 2014 Jun;28(6):1299-307. doi: 10.1038/leu.2013.375. Epub 2013 Dec 17. PMID 24342950
- [Background] Martinez-Lopez J, Lahuerta JJ, Pepin F, Gonzalez M, Barrio S, Ayala R, Puig N, Montalban MA, Paiva B, Weng L, Jimenez C, Sopena M, Moorhead M, Cedena T, Rapado I, Mateos MV, Rosinol L, Oriol A, Blanchard MJ, Martinez R, Blade J, San Miguel J, Faham M, Garcia-Sanz R. Prognostic value of deep sequencing method for minimal residual disease detection in multiple myeloma. Blood. 2014 May 15;123(20):3073-9. doi: 10.1182/blood-2014-01-550020. Epub 2014 Mar 19. PMID 24646471
- [Background] Uniform requirements for manuscripts submitted to biomedical journals: Writing and editing for biomedical publication. J Pharmacol Pharmacother. 2010 Jan;1(1):42-58. No abstract available. PMID 21808590